CLINICAL TRIAL: NCT02771028
Title: A Randomized Wait-list Controlled Trial on the Use of Emotional Freedom Techniques as an Intervention Strategy to Reduce Patient Reported Cognitive Complaints in Cancer Survivors on Behalf of the Belgian Society for Medical Oncology (BSMO)-Cancer Survivorship Taskforce
Brief Title: Emotional Freedom Techniques to Reduce Patient Reported Cognitive Complaints in Cancer Survivors
Acronym: EMOTICON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); AZ Klina (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Medical Oncologist, General Hospital Groeninge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AZGS2016034
Record Dates: First submitted 2016-04-21; First posted 2016-05-12 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Subjective Cognitive Complaints; Cancer
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Intervention group (Experimental): Patients assigned to intervention group receive an 8-week EFT-program
  Interventions: Behavioral: Emotional Freedom Techniques
- Control group (No Intervention): Patients assigned to control group are placed on a waitlist for a period of 8 weeks

INTERVENTIONS:
Behavioral: Emotional Freedom Techniques
  Arms: Intervention group

SUMMARY:
The aim of this study is to further validate the CDT as a screening tool for identifying elderly cancer patients in need of a more in-depth cognitive evaluation within comprehensive geriatric assessment (CGA) and to validate the pre-defined cut-off score of ≤ 4 according to the Freund scoring system. All geriatric patients that are diagnosed with cancer will be screened by the oncology clinical nurse specialists attached to the respective multi-disciplinary clinics with the VES-13 and G8 questionnaire. Patients that screen positive, will be offered referral to the multi-disciplinary onco-geriatric program where a member of the research team will implement a full geriatric evaluation under supervision of the medical oncologist and/or geriatrician who will then formulate recommendations and might suggest referral to other health care providers. Individual results and survival data of all the patients that have given their informed consent will be registered in a database.

DETAILED DESCRIPTION:
In this trial the investigators aim to establish whether Emotional Freedom Techniques (EFT) can reduce cognitive complaints in cancer survivors. All consenting patients aged 18 years or above, who have been diagnosed with a solid tumour of hematologic malignancy and who have completed or are in the late phase of a chemotherapy, radiotherapy, anti-hormonal or targeted therapy treatment, can participate in this trial. Patients should suffer from subjective cognitive complaints based on a score of 43 or more on the Cognitive Failure Questionnaire (CFQ). These patients will be randomly assigned to either the control or intervention group. Patients in the intervention group will be scheduled to receive an 8-week EFT intervention program. Other patients will be placed on an 8-week wait list after which patients will also start the EFT program.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached a minimum age of 18 years at the time of enrolment
* Histologically confirmed diagnosis of a solid cancer or hematologic malignancy
* Patients should have received chemo- or radiotherapy, targeted therapy of hormonal treatment before enrollment (active treatment with anti-hormonal therapy or brachytherapy is allowed)
* Patients can be included in the latest phase of their chemotherapy, radiotherapy, anti-hormonal or targeted therapy treatment
* Patients should have been treated with curative intent or have an expected life expectancy of at least 5 years
* Patients must suffer from subjective cognitive complaints based on the Cognitive Failure Questionnaire (cut-off ≥ 43)
* Patients should be able to adequately communicate in Dutch or French
* Patients should present with a sufficient mental and physical functional status (according to investigator's judgment)

Exclusion Criteria:

* Patients who received a treatment with palliative intent
* Patients showing signs of mental deterioration
* Patients suffering from an organic brain syndrome
* Patients who are alcohol or drug dependent
* Patients with a major psychiatric or neurologic disorder that could potentially invalidate assessment; a prior or current diagnosis of a depressive, anxiety or adjustment disorder is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2016-10-01; Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in cognitive complaints measured by Cognitive Failure Questionnaire | Week 8, 16, 24
  Score of <43 on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome

SECONDARY OUTCOMES:
Change in fatigue measured by Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale | Week 8, 16, 24
  Reduction in score on FACIT Fatigue scale ; Minimum value: 0; Maximum value: 52; Higher scores mean worse outcome
Change in psychological distress measured by Distress Thermometer | Week 8, 16, 24
  Reduction in the score on the Distress Thermometer ; Minimum value: 0; Maximum value: 10; Higher scores mean worse outcome
Change in depressive symptoms measured by Beck Depression Inventory II | Week 8, 16, 24
  Reduction in score on Beck Depression Inventory II ; Minimum value: 0; Maximum value: 63; Higher scores mean worse outcome
Change in quality of life measured by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 | Week 8, 16, 24
  Improvement of the scores on the Global Health scale, functional scale and symptom scale ; Minimum value: 30; Maximum value: 126; Higher scores mean better outcome
Chang in quality of life measured by EQ-5D-3L | Week 8, 16, 24
  Improvement on the score on the EQ-5D-3L; Minimum value: -0.285; Maximum value: 1; Higher scores mean better outcome
Change in long-term quality of life measured by the EuroQol EQ-5D-3L | 6 months and 12 months
  Improvement on the score on the EQ-5D-3L; Minimum value: -0.285; Maximum value: 1; Higher scores mean better outcome
Number of cancer survivors presenting with cognitive complaints as measured by Cognitive Failure Questionnaire | Week 8, 16, 24
  Number of cancer survivors presenting with cognitive complaints as measured by Cognitive Failure Questionnaire
Influence of age on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of age and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of gender on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of gender and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of distress on cognitive complaints in cancer survivors as measured by Distress Thermometer | Week 8, 16, 24
  Interaction effect of distress and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of fatigue (FACIT-Fatigue Scale) on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of fatigue and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of cancer type on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of cancer type and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of cancer stage on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of cancer stage and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire
Influence of the received treatment on cognitive complaints in cancer survivors | Week 8, 16, 24
  Interaction effect of treatment and score on the Cognitive Failure Questionnaire ; Minimum value: 0; Maximum value: 100; Higher scores mean worse outcome; cut-off at score of 43 on the Cognitive Failure Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD, PhD, MSc, FRCP, Principal Investigator — AZ Groeninge
Locations (3):
- Belgium (3):
  - General Hospital Klina Brasschaat, Brasschaat
  - Brussels University Hospital, Brussels
  - General Hospital Groeninge, Kortrijk

REFERENCES:
- [Derived] Tack L, Lefebvre T, Lycke M, Langenaeken C, Fontaine C, Borms M, Hanssens M, Knops C, Meryck K, Boterberg T, Pottel H, Schofield P, Debruyne PR. A randomised wait-list controlled trial to evaluate Emotional Freedom Techniques for self-reported cancer-related cognitive impairment in cancer survivors (EMOTICON). EClinicalMedicine. 2021 Aug 19;39:101081. doi: 10.1016/j.eclinm.2021.101081. eCollection 2021 Sep. PMID 34466793